CLINICAL TRIAL: NCT02333617
Title: Manual Therapy to Treat Gluteus Medius Trigger Points to Improve Hip Abduction Strength in Patients With Anterior Knee Pain.
Brief Title: Manual Therapy to Treat Gluteus Medius Trigger Points
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Mitchell Selhorst (Other)
Responsible Party: Sponsor-Investigator, Mitchell Selhorst, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB14-00621
Record Dates: First submitted 2014-12-23; First posted 2015-01-07 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Anterior Knee Pain Syndrome; Patellofemoral Pain Syndrome
Keywords: Manual Therapy; Physical Therapy; Dry Needling; Gluteus Medius
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Dry Needling; Papaverine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dry Needling and Exercise (Experimental): Dry Needling to treat gluteus medius trigger points followed by hip and core exercises.
  Interventions: Other: Dry Needling; Other: Hip and core strengthening exercises
- Soft Tissue Mobilization (Active Comparator): Soft tissue mobilization to treat gluteus medius trigger points followed by hip and core exercises.
  Interventions: Other: Soft Tissue Mobilization; Other: Hip and core strengthening exercises
- Placebo Control (Placebo Comparator): Placebo to control for hands on time and attention from therapist followed by hip and core exercises.
  Interventions: Other: Placebo Control; Other: Hip and core strengthening exercises

INTERVENTIONS:
Other: Dry Needling — Dry Needling will be performed on the patient's ipsilateral gluteus medius muscle with the patient in sidelying. The treating therapist will use the appropriate needle based upon patient's size and location of trigger point [No. 5 (0.25 x 40mm), No. 8 (0.30 x 50mm), or No. 11 (0.30 x 75mm)]. They will target trigger points identified in the ipsilateral gluteus medius. Once the needling is inserted into the trigger point the needle will be moved in multiple directions until the first local twitch response is noted. Once the first local twitch response is obtained, the needling will be performed in an up-and-down fashion, performing 2- to 3-mm vertical motions with no rotations (fast-in and fast-out technique), at approximately 1 Hz for 25 to 30 seconds, with the aim of eliciting local twitch responses. The treating therapist can dry needle each trigger point identified in the gluteus medius with a maximum treatment time of 5 minutes.
  Arms: Dry Needling and Exercise
Other: Soft Tissue Mobilization — Soft tissue mobilization will be performed on the patient's ipsilateral gluteus medius muscle with the patient in sidelying. The treating therapist will apply firm pressure with the palm and side of their hand. The treating therapist will mobilize the gluteus medius muscle in 4 separate directions (Proximal-Distal, Distal-Proximal, Medial-Lateral, and Lateral-Medial). The treating therapist will apply the pressure to reach the upper limit of the patient's tolerable discomfort. At any point in time the patient can request for the therapist to decrease the pressure applied. The treating therapist will perform soft tissue mobilization for 20 mobilizing strokes in each of the 4 directions.
  Arms: Soft Tissue Mobilization
Other: Placebo Control — Treating therapist will place hands on the patient's gluteus medius muscle and gently rub, but not apply enough pressure to treat the muscles trigger point. This placebo control is designed to account for hands on time from therapist in the 2 other treatment groups, as well as blinding patient to treatment group.
  Arms: Placebo Control
Other: Hip and core strengthening exercises — Patient will perform standardized hip and core exercises using body weight, and elastic bands for resistance. Exercises will take approximately 40 minutes to complete.

SUMMARY:
This is a blinded randomized controlled trial to assess the effectiveness of manual therapy to improve hip abduction strength in patients with acute anterior knee pain.

The primary objective of this study is to see if manual therapy to the gluteus medius can significantly alter within-session measurements of hip abductor strength in patients with anterior knee pain.

The secondary objective of this study is to see if manual therapy to the gluteus medius can significantly alter within session pain in patients with anterior knee pain.

DETAILED DESCRIPTION:
People with anterior knee pain have significant hip abductor muscle weakness compared to healthy people (Prins, 2009). Hip abductor weakness has a strong correlation with impaired lower extremity mechanics and increased pain with functional activity (Stickler et al. 2014). A study by Roach et al in 2013 found that 97% of patients with anterior knee pain had a trigger point in their gluteus medius muscle, while only 23% of healthy controls had trigger points. Trigger points alter normal muscle activity and increase pain in patients (Lucas, 2010, Ibarra et al 2011). Hip abduction strengthening has been found to significantly decrease pain and improve function in patients with anterior knee pain (Earl, 2011). By decreasing trigger points in the gluteus medius the investigators may be able to increase hip abduction strength reducing pain and dysfunction in patients with anterior knee pain.

Both Dry Needling (DN) and Soft Tissue Mobilization (STM) are manual therapy interventions commonly used by physical therapist to decrease trigger points in muscles. Currently, no research has examined the effectiveness of manual therapy to treat trigger points and improve hip abductor strength in patients with anterior knee pain. Clinically, the investigators have noted that after a patient has been treated with STM or DN that the investigators see immediate improvements in hip abduction strength. The investigators do not know if noted improvements result from repeated strength testing practice or actual improved firing strength of muscles.

The primary objective of this study is to see if manual therapy to the gluteus medius can significantly alter within-session measurements of hip abductor strength in patients with anterior knee pain.

The secondary objective of this study is to see if manual therapy to the gluteus medius can significantly alter within session pain in patients with anterior knee pain.

Patients referred to our physical therapy clinic for anterior knee pain will be considered for this study. After explaining the study and answering any patient or parent questions, informed consent will be obtained for those individuals wishing to participate. The participants will be screened to see if they meet the inclusion criteria, and will be randomly to a treatment group (Dry Needling, Soft Tissue Mobilization, Placebo control). This will be a single blinded research study with the assessor being blinded to the intervention. The therapist who performs the hip abductor strength measurements will not be the same therapist who performs the experimental interventions. The patient cannot be blinded to the treatment that they receive. The therapist performing the intervention will open a sealed envelope that allocates patient to Dry Needling, Soft Tissue Mobilization, or Sham Needling group. Following the experimental intervention all patients will perform the same hip and core exercise protocol.

Pre-treatment evaluation measures will be taken on the patient blinded assessor.

These will consist of:

* Hand held dynamometer hip abduction strength measurements.
* Pain with single leg squat

The subject will then receive the appropriate treatment based on his/her random assignment to experimental treatment groups by the treating therapist.

Post-treatment evaluation measures will be taken on all patients by the blinded assessor immediately following treatment. These will be the same measures taken pre-treatment.

* Hand held dynamometer hip abduction strength measurements.
* Pain with single leg squat Patients will then perform the same hip and core exercise protocol, Following these exercises Post-Exercise evaluation measures by the blinded assessor. These will be the same measures taken pre-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Acute anterior knee pain of <90days
* Ipsilateral hip abductor weakness of >15%

  * 2/10 pain with single leg squat

Exclusion Criteria:

* Contraindication to dry needling or soft tissue mobilization
* Non-mechanical anterior knee pain
* Fear of needles

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in Hip Abduction Dynamometer test | Baseline,Immediately Post-Intervention (anticipated at 5 minutes after baseline testing), Immediately Post-Execise (anticipated to be 1 hour after baseline testing)
  Isometric maximal voluntary contraction strength of the hip abductor muscles will be measured with a portable dynamometer. The dynamometer is placed so as the testing pad is positioned 5cm proximal to the lateral femoral condyle.
  Two to three maximal voluntary contraction trials will be permitted. The subjects will be instructed to produce their maximal force without any concern for the rate of force development. The duration of these contractions will be 5 seconds, and thirty seconds of rest will be given between trials. A third trial is completed only if the difference between the first two maximal voluntary contractions is >10%.
  • Hip abduction strength will be expressed as a percentage of the patient body weight.

SECONDARY OUTCOMES:
Change in Numeric Pain Rating Scale (NPRS) during single leg squat | Baseline,Immediately Post-Intervention (anticipated at 5 minutes after baseline testing), Immediately Post-Execise (anticipated to be 1 hour after baseline testing)
  * Patients will perform 5 single leg squats with the tested limb being the stance limb. Patient will keep hands on their hips and are encouraged to keep their hips level and the center of their knee in line with their second toe during the squat.
  * Patient will be asked to rate their highest pain during the Single Leg squat test using the Numeric Pain Rating Scale (NPRS). The NPRS is an 11-point pain-rating scale ranging from 0 (no pain) to 10 (worst imaginable pain) to assess highest pain intensity during the single leg squat test.
  A change of 2 points on the NPRS has been found to be the minimal clinically important difference found previously in research ( Childs, 2005)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Selhorst, DPT, Principal Investigator — Nationwide Childrens Hospital
Locations (1):
- Nationwide Children's Hospital Sports and Ortho PT East Broad, Columbus, Ohio, United States

REFERENCES:
- [Background] Ireland ML, Willson JD, Ballantyne BT, Davis IM. Hip strength in females with and without patellofemoral pain. J Orthop Sports Phys Ther. 2003 Nov;33(11):671-6. doi: 10.2519/jospt.2003.33.11.671. PMID 14669962
- [Background] McCurdy K, Walker J, Armstrong R, Langford G. Relationship between selected measures of strength and hip and knee excursion during unilateral and bilateral landings in women. J Strength Cond Res. 2014 Sep;28(9):2429-36. doi: 10.1519/JSC.0000000000000583. PMID 24942172
- [Background] Munro A, Herrington L, Carolan M. Reliability of 2-dimensional video assessment of frontal-plane dynamic knee valgus during common athletic screening tasks. J Sport Rehabil. 2012 Feb;21(1):7-11. doi: 10.1123/jsr.21.1.7. Epub 2011 Nov 15. PMID 22104115
- [Background] Hua NK, Van der Does E. The occurrence and inter-rater reliability of myofascial trigger points in the quadratus lumborum and gluteus medius: a prospective study in non-specific low back pain patients and controls in general practice. Pain. 1994 Sep;58(3):317-323. doi: 10.1016/0304-3959(94)90125-2. PMID 7838580
- [Background] Prins MR, van der Wurff P. Females with patellofemoral pain syndrome have weak hip muscles: a systematic review. Aust J Physiother. 2009;55(1):9-15. doi: 10.1016/s0004-9514(09)70055-8. PMID 19226237
- [Background] Roach S, Sorenson E, Headley B, San Juan JG. Prevalence of myofascial trigger points in the hip in patellofemoral pain. Arch Phys Med Rehabil. 2013 Mar;94(3):522-6. doi: 10.1016/j.apmr.2012.10.022. Epub 2012 Nov 2. PMID 23127304
- [Background] Schmidt J, Iverson J, Brown S, Thompson PA. Comparative reliability of the make and break tests for hip abduction assessment. Physiother Theory Pract. 2013 Nov;29(8):648-57. doi: 10.3109/09593985.2013.782518. Epub 2013 May 24. PMID 23706084
- [Background] Stickler L, Finley M, Gulgin H. Relationship between hip and core strength and frontal plane alignment during a single leg squat. Phys Ther Sport. 2015 Feb;16(1):66-71. doi: 10.1016/j.ptsp.2014.05.002. Epub 2014 Jun 3. PMID 25070759
- [Background] Thorborg K, Petersen J, Magnusson SP, Holmich P. Clinical assessment of hip strength using a hand-held dynamometer is reliable. Scand J Med Sci Sports. 2010 Jun;20(3):493-501. doi: 10.1111/j.1600-0838.2009.00958.x. Epub 2009 Jun 23. PMID 19558384
- [Background] Widler KS, Glatthorn JF, Bizzini M, Impellizzeri FM, Munzinger U, Leunig M, Maffiuletti NA. Assessment of hip abductor muscle strength. A validity and reliability study. J Bone Joint Surg Am. 2009 Nov;91(11):2666-72. doi: 10.2106/JBJS.H.01119. PMID 19884441
- [Background] Beenakker EA, van der Hoeven JH, Fock JM, Maurits NM. Reference values of maximum isometric muscle force obtained in 270 children aged 4-16 years by hand-held dynamometry. Neuromuscul Disord. 2001 Jul;11(5):441-6. doi: 10.1016/s0960-8966(01)00193-6. PMID 11404114
- [Background] Bohannon RW. Reference values for extremity muscle strength obtained by hand-held dynamometry from adults aged 20 to 79 years. Arch Phys Med Rehabil. 1997 Jan;78(1):26-32. doi: 10.1016/s0003-9993(97)90005-8. PMID 9014953
- [Background] Crossley KM, Zhang WJ, Schache AG, Bryant A, Cowan SM. Performance on the single-leg squat task indicates hip abductor muscle function. Am J Sports Med. 2011 Apr;39(4):866-73. doi: 10.1177/0363546510395456. Epub 2011 Feb 18. PMID 21335344
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561